CLINICAL TRIAL: NCT02778529
Title: Insights Into Impaired Arm Motor Control on Bilateral and Unilateral Functional Activities After Injury: A Kinematic Study
Brief Title: Arm Motor Control on Bi and Uni ADLs
Acronym: BiAs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Equipment Failure
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 820251
Record Dates: First submitted 2016-03-30; First posted 2016-05-20 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Peripheral Neuropathy; Spinal Cord Injuries; Cerebral Palsy
Keywords: stroke; amputees; spinal cord injuries; cerebral palsy; robotics; rehabilitation
MeSH Terms: conditions — Stroke; Peripheral Nervous System Diseases; Spinal Cord Injuries; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Upper Limb Assessment on ADLs (Other): Bilateral assessment robots (BiAS) Evaluate upper limb kinematics of Stroke, Amputees, SCI, Cerebral Palsy and Health Subjects will be assessed as they complete unilateral and bilateral activities of daily living. Subjects will complete exercises in 1 session
  Interventions: Device: Bilateral assessment robots (BiAS)

INTERVENTIONS:
Device: Bilateral assessment robots (BiAS) — The BiAS are two passive desktop robots that will be used in this study to measure right and left arm kinematics for 4 different groups of patients.

SUMMARY:
This study is being performed to assess how certain chronic disabilities - stroke, upper extremity (UE) amputation, spinal cord injuries (SCI), cerebral palsy (CP) - differ from healthy subjects in their ability to perform ADLs. By studying the kinematics of the respective cohort of study participants as they are assessed performing common activities of daily living (ADLS), the investigators research team aims to better understand how impaired neural pathways, and pathways that have been impaired at various points along the pathway, deleteriously affect ADLs in patients with differing long-term disabilities.

DETAILED DESCRIPTION:
Cross-sectional study comparing bilateral ADL activities for stroke survivors, SCI paraplegics, UE amputees, adults with CP, and healthy controls. The study participants will perform 4 ADL tasks with the BiAS passive robots. From these tasks, the BiAS robots will provide information regarding position, velocity, distance, displacement, etc. This, along with video information provided by the 3D Kinect and EEG neuroheadset, will be used as the basis of the investigators data and aid in informing members of the research team on how the respective impairments affected upper limb kinematics on ADL tasks.

Participation in the study will include the following steps:

1. Informed Consent: After arrival, subjects will review and sign the consent form with study personnel present.
2. Pre-Assessments: A member of the research team will evaluate the subjects' upper extremity and assess their ability to use it. Subjects will be evaluated using a battery of assessments such as, but not limited to, the Box and Block, Pin and Prick, and grip strength using a dynamometer.
3. Break: Subjects will be given a 15 minute break.
4. BiAS passive robot system: Subjects will be introduced to the device and each wrist will be placed on to the end of each robot. As common therapy tasks are performed by the subject, the BiAS devices will collect the data along with the video from 3D Kinect, ECG gelled electrodes, and the EEG neuroheadset. After each of the 4 ADL activities, subjects will be asked about their level of exercise and discomfort, if any. After subjects finish all exercises with the BiAS, they will be thanked for their participation in the study.
5. Video and photos may be collected to determine subject quality of ADL movement.

ELIGIBILITY:
Inclusion Criteria:

Study will include subjects 18 years of age or older from any of the below groups:

* Stroke survivors, 3 months post event
* Upper extremity amputees, 3 months post event
* Cervical SCI (C-5 to C-7), 3 months post event
* Cerebral palsy participants
* Healthy participants

Exclusion Criteria:

* The inability to perform at least some aspects of ADL tasks such as drinking, pouring, pinching, and grasping.
* Severe spasticity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Interlimb Coordination | up to 1 week
  Kinematic Variables of Movement Overlap and Phase Difference
Movement Time | up to 1 week
  time to complete a task

SECONDARY OUTCOMES:
Gross Finger Dexterity | up to 1 week
  Box and Block assessment
Sensory Nerve Deficits | up to 1 week
  Pin and Prick assessment
Grip strength | up to 1 week
  Grip Dynamometer measurement of strength
Movement Smoothness | up to 1 week
  Jerkiness on a task

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Johnson, PhD, Principal Investigator — Penn Medicine Rittenhouse
Locations (1):
- Penn Medicine Rittenhouse, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dimwamwa E, Johnson MJ. Kinematic analysis of unilateral and bilateral drinking task after brain and periphery injuries. Annu Int Conf IEEE Eng Med Biol Soc. 2015 Aug;2015:4558-61. doi: 10.1109/EMBC.2015.7319408. PMID 26737308
- [Background] Johnson MJ, Wang S, Bai P, Strachota E, Tchekanov G, Melbye J, McGuire J. Bilateral assessment of functional tasks for robot-assisted therapy applications. Med Biol Eng Comput. 2011 Oct;49(10):1157-71. doi: 10.1007/s11517-011-0817-0. Epub 2011 Sep 1. PMID 21881901